CLINICAL TRIAL: NCT01230151
Title: Sustained Affect of GUIDE (SAGE):A Software Evaluation Study
Brief Title: Feasibility Study to Evaluate Deep Brain Stimulation (DBS) Settings for the Treatment of Parkinson's Disease
Acronym: SAGE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor (Intelect Medical, Inc.) was acquired by Boston Scientific and study was canceled.
Sponsor: Intelect Medical, Inc. (Industry)
Responsible Party: Christopher R. Butson, Ph.D., Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 017-0002
Record Dates: First submitted 2010-10-27; First posted 2010-10-28 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2011-02

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation; DBS; Parkinson's disease; PD; Patients who have a preexisting Deep Brain Stimulation (DBS) system for the treatment of Parkinson's disease (PD)
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical (Active Comparator): Stimulation settings predetermined clinically (Clinical)
  Interventions: Device: Clinically defined stimulation parameters
- Model (Experimental): stimulation settings derived from a patient-specific computer-based model (Model)
  Interventions: Device: GUIDE software, Version 0.1

INTERVENTIONS:
Device: GUIDE software, Version 0.1 — The GUIDE software uses computer-based models to determine the spread of stimulation from DBS therapy into surrounding nuclei of the brain. The software models stimulation and is not used to program or communicate with the patient's implanted DBS System. The software was recently validated in a multi-center clinical study.
  Arms: Model
Device: Clinically defined stimulation parameters — Stimulation parameters clinically determined prior to start of clinical study
  Arms: Clinical

SUMMARY:
The purpose of this study is to assess the cognitive performance in patients with advanced Parkinson's disease receiving Deep Brain Stimulation (DBS) with settings predetermined clinically to settings derived from a patient-specific computational model.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able and willing to provide informed consent to participate in the study.
* The patient's implanted DBS system shall be the Medtronic, Inc. Activa® System. The Medtronic Activa System may consists of either, Soletra®, Kinetra® Activa® RC, or Activa® PC Neurostimulator(s) and two DBS Leads (Model 3387 or 3389).
* Patient shall have bilateral DBS of the subthalamic nucleolus (STN).
* Patient shall have stable DBS stimulation without changes in stimulation parameters for no less than 3 months prior to enrollment.
* Patient shall have stable and optimal regimen of antiparkinson drug therapy for no less than 3 months prior to enrollment.
* Patient, and caregiver if applicable, is able and willing to be available for study visits throughout the duration of the study (e.g. no planned relocation of residence or extended vacation during the study that would prevent compliance with study visit schedule).
* Availability, from the patient's medical records, of a Pre-op MRI and high resolution CT with artifact reduction no less than six (6) weeks post-op.
* Patient shall have Hoehn and Yahr stage III or worse when off stimulation and off medication.
* Patient shall have demonstrated good response to L-DOPA, defined as no less than a 30% improvement in a UPDRS-III motor exam following the administration of L-DOPA during their screening neurological exam.
* Patient shall have demonstrated good response to DBS following the administration of DBS while off medication, defined as an improvement in UPDRS-III motor scores better than their improvement to L-DOPA (as determine in above) or no less than 20% worse of an improvement.

Exclusion Criteria:

* Evidence of secondary or atypical Parkinsonism as suggested by: stroke, encephalitis, exposure to toxins, neuroleptic antipsychotics, neurologic signs of upper motor neuron or cerebellar involvement, or supranuclear palsy.
* Dementia as evidenced by a mini-mental state examination of 24 or below (MMSE ≥ 24).
* Prior participation in the Intelect Medical GUIDE study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
sustained improvement in working memory | 2 Months
  The primary endpoint of this study is to determine whether or not sustained improvement in working memory can be obtained during DBS with stimulation settings derived from a patient-specific computer-based model (Model) as compared with stimulation settings predetermined clinically (Clinical).

SECONDARY OUTCOMES:
Quality of Life (QOL)improvements | 2 Months
  The secondary endpoints will evaluate whether or not sustained cognitive improvements translate into other aspects of the patient's life (e.g. mood, activities of daily living, apathy, etc.) during DBS with stimulation settings derived from a patient-specific computer-based model (Model) as compared with stimulation settings predetermined clinically (Clinical).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of Florida, Gainesville, Florida
  - North Shore University Hospital, Manhasset, New York
  - Evergreen Healthcare, Kirkland, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Frankemolle AM, Wu J, Noecker AM, Voelcker-Rehage C, Ho JC, Vitek JL, McIntyre CC, Alberts JL. Reversing cognitive-motor impairments in Parkinson's disease patients using a computational modelling approach to deep brain stimulation programming. Brain. 2010 Mar;133(Pt 3):746-61. doi: 10.1093/brain/awp315. Epub 2010 Jan 7. PMID 20061324
- See also: Sponsor website — http://www.intelectmedical.com/